CLINICAL TRIAL: NCT03143101
Title: A Phase 4 Double-blind Study to Evaluate the Shedding and Immunogenicity of Trivalent and Quadrivalent Formulations of FluMist in Children 24 to < 48 Months of Age
Brief Title: Evaluate the Shedding and Immunogencity of Different Formulations of FluMist in Children 24 to <48 Months of Age
Acronym: FluMist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D2560C00013
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Influenza; Healthy
Keywords: FluMist Quadrivalent; Trivalent; Influenza; Vaccine; Prevention
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FluMist trivalent (2015-2016) (Experimental): Participants will receive intranasal spray of 0.2 milliliter (mL) (total dose in both nostrils) FluMist trivalent vaccine on Days 1 and 28. Each 0.2 mL dose contained 10^7±0.5 fluorescent focus units (FFU) of each vaccine strain. Strains included in the trivalent vaccine were: A/H1N1 (A/Bolivia/559/2013), A/H3N2 (A/Switzerland/9715293/2013), and B/Phuket/3073/2013 (B/Yamagata-lineage).
  Interventions: Biological: FluMist trivalent (2015-2016)
- FluMist Quadrivalent (2015-2016) (Experimental): Participants will receive intranasal spray of 0.2 mL (total dose in both nostrils) FluMist quadrivalent vaccine on Days 1 and 28. Each 0.2 mL dose contained 10^7±0.5 FFU of each vaccine strain. Strains included in the vaccine were A/H1N1 (A/Bolivia/559/2013), A/H3N2 (A/Switzerland/9715293/2013), B/Phuket/3073/2013 (B/Yamagata-lineage), and B/Brisbane/60/2008 (B/Victoria-lineage).
  Interventions: Biological: FluMist Quadrivalent (2015-2016)
- FluMist Quadrivalent (2017-2018) (Experimental): Participants will receive intranasal spray of 0.2 mL (total dose in both nostrils) FluMist quadrivalent vaccine on Days 1 and 28. Each 0.2 mL dose contained 10^7±0.5 FFU of each vaccine strain. Strains included in the vaccine were the new A/H1N1 (A/Slovenia/2903/2015), A/H3N2 (A/New Caledonia/71/2014), B/Phuket/3073/2013 (B/Yamagata-lineage), and B/Brisbane/60/2008 (B/Victoria-lineage).
  Interventions: Biological: FluMist Quadrivalent (2017-2018)

INTERVENTIONS:
Biological: FluMist trivalent (2015-2016) — 0.2 mL (total dose in both nostrils) on Days 1 and 28. Each 0.2 mL dose will contain 10^7±0.5 FFU of each vaccine strain.
  Arms: FluMist trivalent (2015-2016)
Biological: FluMist Quadrivalent (2015-2016) — 0.2 mL (total dose in both nostrils) on Days 1 and 28. Each 0.2 mL dose will contain 10^7±0.5 FFU of each vaccine strain.
  Arms: FluMist Quadrivalent (2015-2016)
Biological: FluMist Quadrivalent (2017-2018) — 0.2 mL (total dose in both nostrils) on Days 1 and 28. Each 0.2 mL dose will contain 10^7±0.5 FFU of each vaccine strain.
  Arms: FluMist Quadrivalent (2017-2018)

SUMMARY:
This study is being conducted to compare the immunogenicity, safety, and viral shedding of a new A/H1N1 strain that will be incorporated into the FluMist quadrivalent formulation for the 2017-2018 influenza season with the previous A/H1N1 strain that was included in the vaccine in the 2015-2016 influenza season.

DETAILED DESCRIPTION:
This randomized, double-blind, multi-center study will enroll approximately 200 children 24 to less than (<) 48 months of age. Participants will be randomized in a 1:1:1 ratio to receive two doses of either FluMist quadrivalent 2017-2018, FluMist quadrivalent 2015-2016 formulation, or FluMist trivalent 2015-2016 formulation.

Participants will be screened within 30 days prior to randomization. Randomization will be stratified according to whether the participant ever received prior influenza vaccination. Approximately 50% of the participants will not have been previously vaccinated. All participants will receive two doses of investigational product on Study Days 1 and 28, and followed for a 28-day follow-up period after each dose. Blood and nasal samples will be collected and safety evaluations perfomed.

The duration of participants participation is approximately 2 to 3 months. The study will be conducted during the influenza "off-season" in the US. After completion of the study all participants will be offered and strongly encouraged to receive an inactivated influenza vaccine approved for use in the US for the 2017-2018 influenza season.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 24 months to < 48 months of age
* Healthy by medical history and physical examination or presence of stable underlying chronic medical condition for which hospitalization has not been required in the previous year

Key Exclusion Criteria:

* History of allergic disease or reactions likely to be exacerbated by any component of the investigational product
* Acute illness or evidence of significant active infection (including fever >= 100.4 degrees Fahrenheit (38.0 degrees Celsius) at randomization
* History of asthma or history of recurrent wheezing
* Any known immunosuppressive condition or immune deficiency disease
* Current or expected receipt of immunosuppressive medications within a 28 day window around vaccination
* Use of aspirin or salicylate-containing medications within 28 days prior to randomization or expected receipt thru 28 days after vaccination
* Use of antiviral agents with activity against influenza viruses within 48 hours prior to first dose of investigational product or anticipated use of such agents through the end of the study follow-up period
* Receipt of any non-study seasonal influenza vaccine within 90 days of Dose 1 or planned receipt of non-study seasonal influenza vaccine prior to 28 days after last vaccination
* Receipt of immunoglobulin or blood products within 90 days before randomization into the study or expected receipt during study participation
* Known or suspected mitochondrial encephalomyopathy
* History of Guillian-Barre syndrome
* Administration of intranasal medications within 10 days prior to randomization, for expected receipt through 10 days after administration of each dose of investigational product

Ages: 24 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Research Site, Savannah, Georgia
  - Research Site, Bardstown, Kentucky
  - Research Site, St Louis, Missouri
  - Research Site, Norfolk, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Binghamton, New York
  - Research Site, Dakota Dunes, South Dakota
  - Research Site, Fort Worth, Texas
  - Research Site, San Angelo, Texas
  - Research Site, Tomball, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, West Jordan, Utah

REFERENCES:
- See also: CSP in PDF-A — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14608&filename=D2560C00013-clinical-study-protocol-v2-CA_redaction_18SEP18_(RM)_Redacted_PDF-A.pdf
- See also: Statistical Analysis Plan (SAP) in PDF-A — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14608&filename=D2560C00013_Statistical_Analysis_Plan_Final_V1.0_PDF-A.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 08 May 2017 through 29 Sep 2017 in the USA.
Pre-assignment Details: A total of 200 participants were randomized and participated in the study.
Groups:
- FluMist Trivalent (2015-2016): Participants received intranasal spray of 0.2 milliliter (mL) (total dose in both nostrils) FluMist trivalent vaccine on Days 1 and 28. Each 0.2 mL dose contained 10^7±0.5 fluorescent focus units (FFU) of each vaccine strain. Strains included in the trivalent vaccine were: A/H1N1 (A/Bolivia/559/2013), A/H3N2 (A/Switzerland/9715293/2013), and B/Phuket/3073/2013 (B/Yamagata-lineage).
- FluMist Quadrivalent (2015-2016): Participants received intranasal spray of 0.2 mL (total dose in both nostrils) FluMist quadrivalent vaccine on Days 1 and 28. Each 0.2 mL dose contained 10^7±0.5 FFU of each vaccine strain. Strains included in the vaccine were A/H1N1 (A/Bolivia/559/2013), A/H3N2 (A/Switzerland/9715293/2013), B/Phuket/3073/2013 (B/Yamagata-lineage), and B/Brisbane/60/2008 (B/Victoria-lineage).
- FluMist Quadrivalent (2017-2018): Participants received intranasal spray of 0.2 mL (total dose in both nostrils) FluMist quadrivalent vaccine on Days 1 and 28. Each 0.2 mL dose contained 10^7±0.5 FFU of each vaccine strain. Strains included in the vaccine were the new A/H1N1 (A/Slovenia/2903/2015), A/H3N2 (A/New Caledonia/71/2014), B/Phuket/3073/2013 (B/Yamagata-lineage), and B/Brisbane/60/2008 (B/Victoria-lineage).
Period: Overall Study
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Started | 67 | 66 | 67
Completed | 65 | 63 | 67
Not Completed | 2 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any investigational drug.
Groups:
- FluMist Trivalent (2015-2016): Participants received intranasal spray of 0.2 mL (total dose in both nostrils) FluMist trivalent vaccine on Days 1 and 28. Each 0.2 mL dose contained 10^7±0.5 FFU of each vaccine strain. Strains included in the trivalent vaccine were: A/H1N1 (A/Bolivia/559/2013), A/H3N2 (A/Switzerland/9715293/2013), and B/Phuket/3073/2013 (B/Yamagata-lineage).
- Total: Total of all reporting groups
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018) | Total
Number analyzed (Participants) | 67 | 66 | 67 | 200
Age, Continuous [Mean (Standard Deviation); unit: months] — Population: As-treated population included all participants who received any investigational drug.
  months | 35.96 (6.41) | 34.96 (6.78) | 34.94 (6.80) | 35.29 (6.65)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: As-treated population included all participants who received any investigational drug.
  Participants
    Female | 27 | 32 | 35 | 94
    Male | 40 | 34 | 32 | 106
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: As-treated population included all participants who received any investigational drug.
  Participants
    Hispanic or Latino | 11 | 9 | 14 | 34
    Not Hispanic or Latino | 56 | 57 | 53 | 166
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: As-treated population included all participants who received any investigational drug.
  Participants
    American Indian or Alaska Native | 0 | 1 | 0 | 1
    Asian | 1 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 2 | 0 | 1 | 3
    Black or African American | 9 | 9 | 13 | 31
    White | 52 | 55 | 49 | 156
    More than one race | 3 | 1 | 3 | 7
    Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With A/H1N1 Hemagglutination Inhibition (HAI) Antibody Seroconversion Rate at Day 28
Description: Seroconversion rate is defined as at least (>=) 4-fold rise from baseline in A/H1N1 HAI antibody titer. Percentage of participants with >= 4-fold rise in A/H1N1 HAI antibody titer at Day 28 is reported. Comparative statistical analysis was planned only for 'FluMist Quadrivalent (2015-2016)' and 'FluMist Quadrivalent (2017-2018)' arms.
Time Frame: Day 28
Population: Immunogenicity population included all participants in the as-treated population (ATP) who had no major protocol deviations judged to have the potential to interfere with the generation or interpretation of an immune response to investigational product. Here, "N" signifies number of participants analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 60 | 56 | 64
Percentage of participants | 10.0 [3.8 to 20.5] | 5.4 [1.1 to 14.9] | 23.4 [13.8 to 35.7]
Statistical Analysis 1: Comparison: FluMist Quadrivalent (2015-2016) vs FluMist Quadrivalent (2017-2018); Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel — p-value is calculated from the Cochran-Mantel-Haenszel (CMH) test adjusting for the prior influenza vaccination status; Mean Difference (Net) = 18.1, 95% CI 2-sided [4.8 to 30.9]

2. Primary Outcome: Percentage of Participants With A/H3N2 HAI Antibody Seroconversion Rate at Day 28
Description: Seroconversion rate is defined as >= 4-fold rise from baseline in A/H3N2 HAI antibody titer. Percentage of participants with >= 4-fold rise in A/H3N2 HAI antibody titer at Day 28 is reported.
Time Frame: Day 28
Population: Immunogenicity population included all participants in the ATP who had no major protocol deviations judged to have the potential to interfere with the generation or interpretation of an immune response to investigational product. Here, "N" signifies number of participants analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 60 | 56 | 64
Percentage of participants | 51.7 [38.4 to 64.8] | 64.3 [50.4 to 76.6] | 31.3 [20.2 to 44.1]

3. Primary Outcome: Percentage of Participants With B/Yamagata HAI Antibody Seroconversion Rate at Day 28
Description: Seroconversion rate is defined as >= 4-fold rise from baseline in B/Yamagata HAI antibody titer. Percentage of participants with >= 4-fold rise in B/Yamagata HAI antibody titer at Day 28 is reported.
Time Frame: Day 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 60 | 56 | 64
Percentage of participants | 50.0 [36.8 to 63.2] | 42.9 [29.7 to 56.8] | 57.8 [44.8 to 70.1]

4. Primary Outcome: Percentage of Participants With B/Victoria HAI Antibody Seroconversion Rate at Day 28
Description: Seroconversion rate is defined as >= 4-fold rise from baseline in B/Victoria HAI antibody titer. Percentage of participants with >= 4-fold rise in B/Victoria HAI antibody titer at Day 28 is reported.
Time Frame: Day 28
Population: Immunogenicity population. B/Victoria strain was not included in the 'FluMist trivalent (2015-2016)' arm. Here, "N" signifies number of participants analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 0 | 56 | 64
Percentage of participants |  | 14.3 [6.4 to 26.2] | 35.9 [24.3 to 48.9]

5. Primary Outcome: Percentage of Participants With A/H1N1 HAI Antibody Seroconversion Rate at Day 56
Description: Seroconversion rate is defined as >= 4-fold rise from baseline in A/H1N1 HAI antibody titer. Percentage of participants with >= 4-fold rise in A/H1N1 HAI antibody titer at Day 56 is reported. Comparative statistical analysis was planned only for 'FluMist Quadrivalent (2015-2016)' and 'FluMist Quadrivalent (2017-2018)' arms.
Time Frame: Day 56
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 59 | 56 | 62
Percentage of participants | 23.7 [13.6 to 36.6] | 12.5 [5.2 to 24.1] | 45.2 [32.5 to 58.3]
Statistical Analysis 1: Comparison: FluMist Quadrivalent (2015-2016) vs FluMist Quadrivalent (2017-2018); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — p-value is calculated from the CMH test adjusting for the prior influenza vaccination status; Mean Difference (Net) = 32.7, 95% CI 2-sided [14.4 to 47.8]

6. Primary Outcome: Percentage of Participants With A/H3N2 HAI Antibody Seroconversion Rate at Day 56
Description: Seroconversion rate is defined as >= 4-fold rise from baseline in A/H3N2 HAI antibody titer. Percentage of participants with >= 4-fold rise in A/H3N2 HAI antibody titer at Day 56 is reported.
Time Frame: Day 56
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 59 | 56 | 62
Percentage of participants | 54.2 [40.8 to 67.3] | 66.1 [52.2 to 78.2] | 40.3 [28.1 to 53.6]

7. Primary Outcome: Percentage of Participants With B/Yamagata HAI Antibody Seroconversion Rate at Day 56
Description: Seroconversion rate is defined as >= 4-fold rise from baseline in B/Yamagata HAI antibody titer. Percentage of participants with >= 4-fold rise in B/Yamagata HAI antibody titer at Day 56 is reported.
Time Frame: Day 56
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 60 | 56 | 62
Percentage of participants | 50.0 [36.8 to 63.2] | 53.6 [39.7 to 67.0] | 54.8 [41.7 to 67.5]

8. Primary Outcome: Percentage of Participants With B/Victoria HAI Antibody Seroconversion Rate at Day 56
Description: Seroconversion rate is defined as >= 4-fold rise from baseline in B/Victoria HAI antibody titer. Percentage of participants with >= 4-fold rise in B/Victoria HAI antibody titer at Day 56 is reported.
Time Frame: Day 56
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 0 | 56 | 62
Percentage of participants |  | 25.0 [14.4 to 38.4] | 40.3 [28.1 to 53.6]

9. Secondary Outcome: Percentage of Participants Who Shed Vaccine Virus by Formulation, Strain, Dose Number, and Baseline Serostatus as Measured by Quantitative Reverse Transcriptase Polymerase Chain Reaction (qRT-PCR)
Description: Quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) was used to measure viral shedding from the nasopharyngeal swabs. Percentage of participants who shed virus are reported.
Time Frame: Days 2, 3, 4, 5, and 7 after Dose 1 (Day 1 dose) and on Days 2, 4, and 6 after Dose 2 (Day 28 dose)
Population: Immunogenicity population. B/Victoria strain was not included in the 'FluMist trivalent (2015-2016)' arm.
Measure: Number; unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 67 | 66 | 67
Percentage of participants
  A/H1N1/HAI seronegative/Dose 1: number analyzed (Participants) | 30 | 43 | 39
  A/H1N1/HAI seronegative/Dose 1 | 86.7 | 81.4 | 94.9
  A/H1N1/HAI seronegative/Dose 2: number analyzed (Participants) | 29 | 43 | 39
  A/H1N1/HAI seronegative/Dose 2 | 17.2 | 25.6 | 46.2
  A/H1N1/HAI seropositive/Dose 1: number analyzed (Participants) | 36 | 22 | 28
  A/H1N1/HAI seropositive/Dose 1 | 86.1 | 63.6 | 71.4
  A/H1N1/HAI seropositive/Dose 2: number analyzed (Participants) | 35 | 21 | 27
  A/H1N1/HAI seropositive/Dose 2 | 22.9 | 23.8 | 29.6
  A/H3N2/HAI seronegative/Dose 1: number analyzed (Participants) | 21 | 35 | 24
  A/H3N2/HAI seronegative/Dose 1 | 100.0 | 100.0 | 95.8
  A/H3N2/HAI seronegative/Dose 2: number analyzed (Participants) | 20 | 35 | 24
  A/H3N2/HAI seronegative/Dose 2 | 55.0 | 60.0 | 79.2
  A/H3N2/HAI seropositive/Dose 1: number analyzed (Participants) | 45 | 30 | 43
  A/H3N2/HAI seropositive/Dose 1 | 95.6 | 83.3 | 95.3
  A/H3N2/HAI seropositive/Dose 2: number analyzed (Participants) | 44 | 29 | 42
  A/H3N2/HAI seropositive/Dose 2 | 47.7 | 44.8 | 59.5
  B/Yamagata/HAI seronegative/Dose 1: number analyzed (Participants) | 51 | 54 | 51
  B/Yamagata/HAI seronegative/Dose 1 | 100.0 | 98.1 | 100.0
  B/Yamagata/HAI seronegative/Dose 2: number analyzed (Participants) | 50 | 53 | 51
  B/Yamagata/HAI seronegative/Dose 2 | 42.0 | 39.6 | 31.4
  B/Yamagata/HAI seropositive/Dose 1: number analyzed (Participants) | 15 | 11 | 16
  B/Yamagata/HAI seropositive/Dose 1 | 73.3 | 81.8 | 93.8
  B/Yamagata/HAI seropositive/Dose 2: number analyzed (Participants) | 14 | 11 | 15
  B/Yamagata/HAI seropositive/Dose 2 | 50.0 | 54.5 | 53.3
  B/Victoria/HAI seronegative/Dose 1: number analyzed (Participants) | 0 | 59 | 39
  B/Victoria/HAI seronegative/Dose 1 |  | 100.0 | 100.0
  B/Victoria/HAI seronegative/Dose 2: number analyzed (Participants) | 0 | 58 | 39
  B/Victoria/HAI seronegative/Dose 2 |  | 44.8 | 53.8
  B/Victoria/HAI seropositive/Dose 1: number analyzed (Participants) | 0 | 6 | 28
  B/Victoria/HAI seropositive/Dose 1 |  | 83.3 | 100.0
  B/Victoria/HAI seropositive/Dose 2: number analyzed (Participants) | 0 | 6 | 27
  B/Victoria/HAI seropositive/Dose 2 |  | 50.0 | 37.0

10. Secondary Outcome: Number of Days of Vaccine Virus Shedding by Formulation, Strain, Dose Number, and Baseline Serostatus as Measured by qRT-PCR
Description: Quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) was used to measure viral shedding from the nasopharyngeal swabs. Number of days of virus shedding are reported.
Time Frame: Days 2, 3, 4, 5, and 7 after Dose 1 (Day 1 dose) and on Days 2, 4 and 6 after Dose 2 (Day 28 dose)
Population: Participants included in immunogenicity population and who shed vaccine virus were analyzed for this outcome measure. B/Victoria strain was not included in the 'FluMist trivalent (2015-2016)' arm.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 66 | 65 | 67
Days
  A/H1N1/HAI seronegative/Dose 1: number analyzed (Participants) | 26 | 35 | 37
  A/H1N1/HAI seronegative/Dose 1 | 2.2 (1.2) | 2.2 (1.0) | 2.8 (1.3)
  A/H1N1/HAI seronegative/Dose 2: number analyzed (Participants) | 5 | 11 | 18
  A/H1N1/HAI seronegative/Dose 2 | 1.2 (0.4) | 1.4 (0.7) | 1.3 (0.5)
  A/H1N1/HAI seropositive/Dose 1: number analyzed (Participants) | 31 | 14 | 20
  A/H1N1/HAI seropositive/Dose 1 | 2.2 (1.0) | 1.9 (0.7) | 2.0 (1.3)
  A/H1N1/HAI seropositive/Dose 2: number analyzed (Participants) | 8 | 5 | 8
  A/H1N1/HAI seropositive/Dose 2 | 1.1 (0.4) | 1.0 (0.0) | 1.1 (0.4)
  A/H3N2/HAI seronegative/Dose 1: number analyzed (Participants) | 21 | 35 | 23
  A/H3N2/HAI seronegative/Dose 1 | 4.5 (1.0) | 4.5 (0.9) | 3.9 (1.2)
  A/H3N2/HAI seronegative/Dose 2: number analyzed (Participants) | 11 | 21 | 19
  A/H3N2/HAI seronegative/Dose 2 | 1.3 (0.6) | 1.1 (0.4) | 1.7 (0.8)
  A/H3N2/HAI seropositive/Dose 1: number analyzed (Participants) | 43 | 25 | 41
  A/H3N2/HAI seropositive/Dose 1 | 3.8 (1.5) | 3.4 (1.6) | 2.5 (1.4)
  A/H3N2/HAI seropositive/Dose 2: number analyzed (Participants) | 21 | 13 | 25
  A/H3N2/HAI seropositive/Dose 2 | 1.3 (0.6) | 1.5 (0.8) | 1.4 (0.6)
  B/Yamagata/HAI seronegative/Dose 1: number analyzed (Participants) | 51 | 53 | 51
  B/Yamagata/HAI seronegative/Dose 1 | 3.6 (1.3) | 3.6 (1.3) | 4.0 (1.1)
  B/Yamagata/HAI seronegative/Dose 2: number analyzed (Participants) | 21 | 21 | 16
  B/Yamagata/HAI seronegative/Dose 2 | 1.3 (0.6) | 1.3 (0.7) | 1.1 (0.3)
  B/Yamagata/HAI seropositive/Dose 1: number analyzed (Participants) | 11 | 9 | 15
  B/Yamagata/HAI seropositive/Dose 1 | 2.5 (1.2) | 3.3 (1.0) | 3.1 (1.6)
  B/Yamagata/HAI seropositive/Dose 2: number analyzed (Participants) | 7 | 6 | 8
  B/Yamagata/HAI seropositive/Dose 2 | 1.1 (0.4) | 1.0 (0.0) | 1.3 (0.5)
  B/Victoria/HAI seronegative/Dose 1: number analyzed (Participants) | 0 | 59 | 39
  B/Victoria/HAI seronegative/Dose 1 |  | 3.9 (1.2) | 4.6 (0.8)
  B/Victoria/HAI seronegative/Dose 2: number analyzed (Participants) | 0 | 26 | 21
  B/Victoria/HAI seronegative/Dose 2 |  | 1.4 (0.6) | 1.4 (0.6)
  B/Victoria/HAI seropositive/Dose 1: number analyzed (Participants) | 0 | 5 | 28
  B/Victoria/HAI seropositive/Dose 1 |  | 2.0 (1.0) | 3.5 (1.5)
  B/Victoria/HAI seropositive/Dose 2: number analyzed (Participants) | 0 | 3 | 10
  B/Victoria/HAI seropositive/Dose 2 |  | 1.0 (0.0) | 1.1 (0.3)

11. Secondary Outcome: Viral Titer by Day, Strain, Dose Number, and Baseline Serostatus as Measured by qRT-PCR
Description: Quantitative reverse transcriptase polymerase chain reaction (qRT-PCR) was used to measure viral titer from the nasopharyngeal swabs. Viral titers are reported.
Time Frame: Day (D) 2, D3, D4, D5, and D7 after Dose 1 (D1 dose) and on D2, D4 and D6 after Dose 2 (D28 dose)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: log10 viral particles/mL
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 66 | 65 | 67
log10 viral particles/mL
  A/H1N1/HAI seronegative/Dose1D2: number analyzed (Participants) | 13 | 16 | 16
  A/H1N1/HAI seronegative/Dose1D2 | 3.79 (0.56) | 3.76 (0.71) | 3.70 (0.49)
  A/H1N1/HAI seronegative/Dose1D3: number analyzed (Participants) | 16 | 20 | 25
  A/H1N1/HAI seronegative/Dose1D3 | 3.66 (0.55) | 3.81 (0.83) | 4.21 (0.97)
  A/H1N1/HAI seronegative/Dose1D4: number analyzed (Participants) | 4 | 6 | 19
  A/H1N1/HAI seronegative/Dose1D4 | 3.63 (0.34) | 3.34 (0.56) | 3.81 (0.94)
  A/H1N1/HAI seronegative/Dose1D5: number analyzed (Participants) | 3 | 3 | 9
  A/H1N1/HAI seronegative/Dose1D5 | 3.12 (0.16) | 3.17 (0.10) | 3.85 (0.48)
  A/H1N1/HAI seronegative/Dose1D7: number analyzed (Participants) | 2 | 0 | 3
  A/H1N1/HAI seronegative/Dose1D7 | 3.17 (0.40) |  | 2.93 (0.23)
  A/H1N1/HAI seronegative/Dose2D2: number analyzed (Participants) | 4 | 7 | 6
  A/H1N1/HAI seronegative/Dose2D2 | 3.68 (0.88) | 3.29 (0.30) | 3.90 (1.04)
  A/H1N1/HAI seronegative/Dose2D4: number analyzed (Participants) | 0 | 3 | 4
  A/H1N1/HAI seronegative/Dose2D4 |  | 3.49 (0.37) | 4.02 (1.24)
  A/H1N1/HAI seronegative/Dose2D6: number analyzed (Participants) | 0 | 0 | 0
  A/H1N1/HAI seropositive/Dose1D2: number analyzed (Participants) | 17 | 9 | 13
  A/H1N1/HAI seropositive/Dose1D2 | 3.66 (0.46) | 3.48 (0.62) | 3.14 (0.45)
  A/H1N1/HAI seropositive/Dose1D3: number analyzed (Participants) | 17 | 7 | 7
  A/H1N1/HAI seropositive/Dose1D3 | 3.39 (0.57) | 4.03 (0.91) | 3.99 (0.84)
  A/H1N1/HAI seropositive/Dose1D4: number analyzed (Participants) | 5 | 2 | 6
  A/H1N1/HAI seropositive/Dose1D4 | 3.09 (0.62) | 3.39 (0.25) | 3.97 (0.73)
  A/H1N1/HAI seropositive/Dose1D5: number analyzed (Participants) | 3 | 0 | 3
  A/H1N1/HAI seropositive/Dose1D5 | 3.35 (0.64) |  | 3.73 (0.62)
  A/H1N1/HAI seropositive/Dose1D7: number analyzed (Participants) | 1 | 0 | 0
  A/H1N1/HAI seropositive/Dose1D7 | 3.10 (NA) — Standard deviation (SD) data not applicable as only one participant was evaluable for this reporting group. |  |
  A/H1N1/HAI seropositive/Dose2D2: number analyzed (Participants) | 6 | 1 | 5
  A/H1N1/HAI seropositive/Dose2D2 | 3.38 (0.78) | 2.86 (NA) — SD data not applicable as only one participant was evaluable for this reporting group. | 3.36 (0.56)
  A/H1N1/HAI seropositive/Dose2D4: number analyzed (Participants) | 0 | 0 | 1
  A/H1N1/HAI seropositive/Dose2D4 |  |  | 3.65 (NA) — SD data not applicable as only one participant was evaluable for this reporting group.
  A/H1N1/HAI seropositive/Dose2D6: number analyzed (Participants) | 0 | 0 | 0
  A/H3N2/HAI seronegative/Dose1D2: number analyzed (Participants) | 19 | 29 | 15
  A/H3N2/HAI seronegative/Dose1D2 | 4.20 (0.99) | 4.15 (0.93) | 3.52 (0.77)
  A/H3N2/HAI seronegative/Dose1D3: number analyzed (Participants) | 19 | 30 | 18
  A/H3N2/HAI seronegative/Dose1D3 | 5.20 (1.12) | 5.39 (1.19) | 4.34 (0.86)
  A/H3N2/HAI seronegative/Dose1D4: number analyzed (Participants) | 20 | 33 | 18
  A/H3N2/HAI seronegative/Dose1D4 | 4.86 (0.99) | 4.51 (1.14) | 4.51 (1.05)
  A/H3N2/HAI seronegative/Dose1D5: number analyzed (Participants) | 18 | 31 | 17
  A/H3N2/HAI seronegative/Dose1D5 | 4.04 (1.09) | 4.16 (1.20) | 3.67 (1.06)
  A/H3N2/HAI seronegative/Dose1D7: number analyzed (Participants) | 14 | 24 | 9
  A/H3N2/HAI seronegative/Dose1D7 | 4.10 (0.97) | 4.12 (0.88) | 3.58 (1.26)
  A/H3N2/HAI seronegative/Dose2D2: number analyzed (Participants) | 7 | 12 | 12
  A/H3N2/HAI seronegative/Dose2D2 | 3.67 (1.03) | 3.33 (0.67) | 3.01 (0.49)
  A/H3N2/HAI seronegative/Dose2D4: number analyzed (Participants) | 0 | 2 | 8
  A/H3N2/HAI seronegative/Dose2D4 |  | 3.41 (0.26) | 3.68 (0.70)
  A/H3N2/HAI seronegative/Dose2D6: number analyzed (Participants) | 0 | 1 | 3
  A/H3N2/HAI seronegative/Dose2D6 |  | 2.72 (NA) — SD data not applicable as only one participant was evaluable for this reporting group. | 3.05 (0.61)
  A/H3N2/HAI seropositive/Dose1D2: number analyzed (Participants) | 38 | 18 | 28
  A/H3N2/HAI seropositive/Dose1D2 | 3.80 (1.07) | 3.98 (1.02) | 3.19 (0.67)
  A/H3N2/HAI seropositive/Dose1D3: number analyzed (Participants) | 33 | 16 | 17
  A/H3N2/HAI seropositive/Dose1D3 | 4.79 (1.29) | 5.06 (1.20) | 3.54 (0.98)
  A/H3N2/HAI seropositive/Dose1D4: number analyzed (Participants) | 31 | 17 | 14
  A/H3N2/HAI seropositive/Dose1D4 | 4.34 (1.03) | 4.45 (1.14) | 4.00 (1.24)
  A/H3N2/HAI seropositive/Dose1D5: number analyzed (Participants) | 26 | 11 | 13
  A/H3N2/HAI seropositive/Dose1D5 | 3.99 (1.05) | 4.01 (0.98) | 3.98 (0.72)
  A/H3N2/HAI seropositive/Dose1D7: number analyzed (Participants) | 21 | 5 | 6
  A/H3N2/HAI seropositive/Dose1D7 | 3.92 (1.06) | 4.10 (1.36) | 3.30 (0.55)
  A/H3N2/HAI seropositive/Dose2D2: number analyzed (Participants) | 16 | 9 | 9
  A/H3N2/HAI seropositive/Dose2D2 | 3.30 (0.89) | 3.55 (0.93) | 3.54 (0.78)
  A/H3N2/HAI seropositive/Dose2D4: number analyzed (Participants) | 3 | 4 | 4
  A/H3N2/HAI seropositive/Dose2D4 | 2.71 (0.62) | 3.38 (0.90) | 3.26 (0.60)
  A/H3N2/HAI seropositive/Dose2D6: number analyzed (Participants) | 1 | 1 | 1
  A/H3N2/HAI seropositive/Dose2D6 | 3.82 (NA) — SD data not applicable as only one participant was evaluable for this reporting group. | 2.32 (NA) — SD data not applicable as only one participant was evaluable for this reporting group. | 3.17 (NA) — SD data not applicable as only one participant was evaluable for this reporting group.
  B/Yamagata/HAI seronegative/Dose1D2: number analyzed (Participants) | 18 | 20 | 21
  B/Yamagata/HAI seronegative/Dose1D2 | 3.93 (0.40) | 4.09 (0.53) | 4.16 (0.58)
  B/Yamagata/HAI seronegative/Dose1D3: number analyzed (Participants) | 26 | 29 | 29
  B/Yamagata/HAI seronegative/Dose1D3 | 4.10 (0.60) | 4.60 (0.77) | 4.72 (0.92)
  B/Yamagata/HAI seronegative/Dose1D4: number analyzed (Participants) | 27 | 29 | 33
  B/Yamagata/HAI seronegative/Dose1D4 | 4.04 (0.61) | 4.60 (0.83) | 4.72 (0.88)
  B/Yamagata/HAI seronegative/Dose1D5: number analyzed (Participants) | 19 | 22 | 29
  B/Yamagata/HAI seronegative/Dose1D5 | 4.56 (0.53) | 4.42 (0.72) | 4.59 (0.80)
  B/Yamagata/HAI seronegative/Dose1D7: number analyzed (Participants) | 19 | 14 | 23
  B/Yamagata/HAI seronegative/Dose1D7 | 4.37 (0.86) | 3.93 (0.50) | 3.98 (0.62)
  B/Yamagata/HAI seronegative/Dose2D2: number analyzed (Participants) | 4 | 5 | 5
  B/Yamagata/HAI seronegative/Dose2D2 | 3.92 (0.31) | 4.10 (0.55) | 3.80 (0.35)
  B/Yamagata/HAI seronegative/Dose2D4: number analyzed (Participants) | 4 | 5 | 0
  B/Yamagata/HAI seronegative/Dose2D4 | 3.74 (0.60) | 3.85 (0.52) |
  B/Yamagata/HAI seronegative/Dose2D6: number analyzed (Participants) | 2 | 0 | 0
  B/Yamagata/HAI seronegative/Dose2D6 | 3.83 (0.35) |  |
  B/Yamagata/HAI seropositive/Dose1D2: number analyzed (Participants) | 3 | 7 | 5
  B/Yamagata/HAI seropositive/Dose1D2 | 3.93 (0.20) | 3.57 (0.19) | 4.15 (0.78)
  B/Yamagata/HAI seropositive/Dose1D3: number analyzed (Participants) | 5 | 6 | 5
  B/Yamagata/HAI seropositive/Dose1D3 | 3.93 (0.58) | 3.92 (0.51) | 4.67 (0.79)
  B/Yamagata/HAI seropositive/Dose1D4: number analyzed (Participants) | 2 | 2 | 7
  B/Yamagata/HAI seropositive/Dose1D4 | 3.46 (0.04) | 4.60 (1.44) | 4.94 (1.28)
  B/Yamagata/HAI seropositive/Dose1D5: number analyzed (Participants) | 1 | 1 | 7
  B/Yamagata/HAI seropositive/Dose1D5 | 3.84 (NA) — SD data not applicable as only one participant was evaluable for this reporting group. | 5.01 (NA) — SD data not applicable as only one participant was evaluable for this reporting group. | 4.82 (0.65)
  B/Yamagata/HAI seropositive/Dose1D7: number analyzed (Participants) | 1 | 0 | 5
  B/Yamagata/HAI seropositive/Dose1D7 | 5.46 (NA) — SD data not applicable as only one participant was evaluable for this reporting group. |  | 3.91 (0.63)
  B/Yamagata/HAI seropositive/Dose2D2: number analyzed (Participants) | 0 | 1 | 3
  B/Yamagata/HAI seropositive/Dose2D2 |  | 3.38 (NA) — SD data not applicable as only one participant was evaluable for this reporting group. | 3.70 (0.11)
  B/Yamagata/HAI seropositive/Dose2D4: number analyzed (Participants) | 0 | 0 | 0
  B/Yamagata/HAI seropositive/Dose2D6: number analyzed (Participants) | 1 | 0 | 0
  B/Yamagata/HAI seropositive/Dose2D6 | 3.92 (NA) — SD data not applicable as only one participant was evaluable for this reporting group. |  |
  B/Victoria/HAI seronegative/Dose1D2: number analyzed (Participants) | 0 | 33 | 25
  B/Victoria/HAI seronegative/Dose1D2 |  | 3.41 (0.58) | 3.49 (0.72)
  B/Victoria/HAI seronegative/Dose1D3: number analyzed (Participants) | 0 | 44 | 31
  B/Victoria/HAI seronegative/Dose1D3 |  | 4.12 (1.02) | 4.39 (0.98)
  B/Victoria/HAI seronegative/Dose1D4: number analyzed (Participants) | 0 | 41 | 35
  B/Victoria/HAI seronegative/Dose1D4 |  | 4.02 (1.13) | 4.58 (1.24)
  B/Victoria/HAI seronegative/Dose1D5: number analyzed (Participants) | 0 | 29 | 34
  B/Victoria/HAI seronegative/Dose1D5 |  | 3.98 (1.05) | 4.09 (1.02)
  B/Victoria/HAI seronegative/Dose1D7: number analyzed (Participants) | 0 | 30 | 26
  B/Victoria/HAI seronegative/Dose1D7 |  | 3.57 (0.79) | 4.14 (0.84)
  B/Victoria/HAI seronegative/Dose2D2: number analyzed (Participants) | 0 | 10 | 6
  B/Victoria/HAI seronegative/Dose2D2 |  | 3.43 (1.01) | 2.94 (0.36)
  B/Victoria/HAI seronegative/Dose2D4: number analyzed (Participants) | 0 | 5 | 3
  B/Victoria/HAI seronegative/Dose2D4 |  | 3.48 (0.88) | 2.67 (0.29)
  B/Victoria/HAI seronegative/Dose2D6: number analyzed (Participants) | 0 | 0 | 0
  B/Victoria/HAI seropositive/Dose1D2: number analyzed (Participants) | 0 | 2 | 11
  B/Victoria/HAI seropositive/Dose1D2 |  | 2.73 (0.01) | 3.10 (0.53)
  B/Victoria/HAI seropositive/Dose1D3: number analyzed (Participants) | 0 | 3 | 14
  B/Victoria/HAI seropositive/Dose1D3 |  | 3.09 (0.42) | 3.96 (1.08)
  B/Victoria/HAI seropositive/Dose1D4: number analyzed (Participants) | 0 | 1 | 16
  B/Victoria/HAI seropositive/Dose1D4 |  | 2.73 (NA) — SD data not applicable as only one participant was evaluable for this reporting group. | 4.40 (0.98)
  B/Victoria/HAI seropositive/Dose1D5: number analyzed (Participants) | 0 | 0 | 15
  B/Victoria/HAI seropositive/Dose1D5 |  |  | 4.26 (0.90)
  B/Victoria/HAI seropositive/Dose1D7: number analyzed (Participants) | 0 | 0 | 12
  B/Victoria/HAI seropositive/Dose1D7 |  |  | 4.00 (0.96)
  B/Victoria/HAI seropositive/Dose2D2: number analyzed (Participants) | 0 | 0 | 4
  B/Victoria/HAI seropositive/Dose2D2 |  |  | 3.41 (0.51)
  B/Victoria/HAI seropositive/Dose2D4: number analyzed (Participants) | 0 | 0 | 0
  B/Victoria/HAI seropositive/Dose2D6: number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Percentage of Participants With Strain-specific Neutralizing Antibody Seroconversion Rates From Baseline Through Days 28 and 56 by Baseline Serostatus
Description: Seroconversion rate is defined as >= 4-fold rise from baseline in strain specific microneutralizing antibody titer. Baseline microneutralization values of less than or equal to (<=) 10 were considered as microneutralization status negative and values greater than (>) 10 were considered microneutralization positive. Percentage of participants with >= 4-fold rise in strain specific neutralizing antibody titer at Days 28 and 56 are reported.
Time Frame: Days 28 and 56
Population: Immunogenicity population. B/Victoria strain was not included in the 'FluMist trivalent (2015-2016)' arm.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 66 | 65 | 67
Percentage of participants
  A/H1N1/Baseline serostatus:negative/Day 28: number analyzed (Participants) | 8 | 20 | 0
  A/H1N1/Baseline serostatus:negative/Day 28 | 0.0 [0.0 to 36.9] | 10.0 [1.2 to 31.7] |
  A/H1N1/Baseline serostatus:negative/Day 56: number analyzed (Participants) | 8 | 20 | 0
  A/H1N1/Baseline serostatus:negative/Day 56 | 37.5 [8.5 to 75.5] | 25.0 [8.7 to 49.1] |
  A/H1N1/Baseline serostatus:positive/Day 28: number analyzed (Participants) | 52 | 36 | 63
  A/H1N1/Baseline serostatus:positive/Day 28 | 3.8 [0.5 to 13.2] | 2.8 [0.1 to 14.5] | 15.9 [7.9 to 27.3]
  A/H1N1/Baseline serostatus:positive/Day 56: number analyzed (Participants) | 51 | 36 | 60
  A/H1N1/Baseline serostatus:positive/Day 56 | 11.8 [4.4 to 23.9] | 2.8 [0.1 to 14.5] | 31.7 [20.3 to 45.0]
  A/H3N2/Baseline serostatus:negative/Day 28: number analyzed (Participants) | 14 | 27 | 15
  A/H3N2/Baseline serostatus:negative/Day 28 | 100.0 [76.8 to 100.0] | 100.0 [87.2 to 100.0] | 46.7 [21.3 to 73.4]
  A/H3N2/Baseline serostatus:negative/Day 56: number analyzed (Participants) | 16 | 26 | 13
  A/H3N2/Baseline serostatus:negative/Day 56 | 93.8 [69.8 to 99.8] | 100.0 [86.8 to 100.0] | 84.6 [54.6 to 98.1]
  A/H3N2/Baseline serostatus:positive/Day 28: number analyzed (Participants) | 46 | 29 | 48
  A/H3N2/Baseline serostatus:positive/Day 28 | 47.8 [32.9 to 63.1] | 34.5 [17.9 to 54.3] | 25.0 [13.6 to 39.6]
  A/H3N2/Baseline serostatus:positive/Day 56: number analyzed (Participants) | 43 | 30 | 47
  A/H3N2/Baseline serostatus:positive/Day 56 | 44.2 [29.1 to 60.1] | 43.3 [25.5 to 62.6] | 14.9 [6.2 to 28.3]
  B/Yamagata/Baseline serostatus:negative/Day 28: number analyzed (Participants) | 44 | 46 | 50
  B/Yamagata/Baseline serostatus:negative/Day 28 | 59.1 [43.2 to 73.7] | 45.7 [30.9 to 61.0] | 58.0 [43.2 to 71.8]
  B/Yamagata/Baseline serostatus:negative/Day 56: number analyzed (Participants) | 44 | 47 | 49
  B/Yamagata/Baseline serostatus:negative/Day 56 | 77.3 [62.2 to 88.5] | 68.1 [52.9 to 80.9] | 75.5 [61.1 to 86.7]
  B/Yamagata/Baseline serostatus:positive/Day 28: number analyzed (Participants) | 16 | 10 | 14
  B/Yamagata/Baseline serostatus:positive/Day 28 | 18.8 [4.0 to 45.6] | 0.0 [0.0 to 30.8] | 14.3 [1.8 to 42.8]
  B/Yamagata/Baseline serostatus:positive/Day 56: number analyzed (Participants) | 16 | 9 | 13
  B/Yamagata/Baseline serostatus:positive/Day 56 | 18.8 [4.0 to 45.6] | 0.0 [0.0 to 33.6] | 7.7 [0.2 to 36.0]
  B/Victoria/Baseline serostatus:negative/Day 28: number analyzed (Participants) | 0 | 48 | 53
  B/Victoria/Baseline serostatus:negative/Day 28 |  | 20.8 [10.5 to 35.0] | 18.9 [9.4 to 32.0]
  B/Victoria/Baseline serostatus:negative/Day 56: number analyzed (Participants) | 0 | 49 | 51
  B/Victoria/Baseline serostatus:negative/Day 56 |  | 16.3 [7.3 to 29.7] | 23.5 [12.8 to 37.5]
  B/Victoria/Baseline serostatus:positive/Day 28: number analyzed (Participants) | 0 | 8 | 10
  B/Victoria/Baseline serostatus:positive/Day 28 |  | 12.5 [0.3 to 52.7] | 10.0 [0.3 to 44.5]
  B/Victoria/Baseline serostatus:positive/Day 56: number analyzed (Participants) | 0 | 7 | 9
  B/Victoria/Baseline serostatus:positive/Day 56 |  | 14.3 [0.4 to 57.9] | 11.1 [0.3 to 48.2]

13. Secondary Outcome: Percentage of Participants With Strain-specific Nasal Immunoglobulin A (IgA) Seroconversion Rate From Baseline Through Days 28 and 56
Description: Seroconversion rate is defined as >= 2-fold rise from baseline in strain speciific nasal IgA antibody titer. Percentage of participants with >= 2-fold rise in strain speciific nasal IgA antibody titer at Days 28 and 56 are reported for this outcome.
Time Frame: Days 28 and 56
Population: Immunogenicity population. B/Victoria strain was not included in the 'FluMist trivalent (2015-2016)' arm.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 66 | 65 | 67
Percentage of participants
  A/H1N1/Day 28: number analyzed (Participants) | 62 | 63 | 67
  A/H1N1/Day 28 | 33.9 [22.3 to 47.0] | 31.7 [20.6 to 44.7] | 40.3 [28.5 to 53.0]
  A/H1N1//Day 56: number analyzed (Participants) | 64 | 60 | 65
  A/H1N1//Day 56 | 40.6 [28.5 to 53.6] | 46.7 [33.7 to 60.0] | 67.7 [54.9 to 78.8]
  A/H3N2//Day 28: number analyzed (Participants) | 63 | 62 | 67
  A/H3N2//Day 28 | 79.4 [67.3 to 88.5] | 79.0 [66.8 to 88.3] | 44.8 [32.6 to 57.4]
  A/H3N2/Day 56: number analyzed (Participants) | 64 | 61 | 65
  A/H3N2/Day 56 | 89.1 [78.8 to 95.5] | 88.5 [77.8 to 95.3] | 55.4 [42.5 to 67.7]
  B/Yamagata//Day 28: number analyzed (Participants) | 63 | 63 | 67
  B/Yamagata//Day 28 | 69.8 [57.0 to 80.8] | 79.4 [67.3 to 88.5] | 77.6 [65.8 to 86.9]
  B/Yamagata//Day 56: number analyzed (Participants) | 64 | 61 | 66
  B/Yamagata//Day 56 | 81.3 [69.5 to 89.9] | 88.5 [77.8 to 95.3] | 86.4 [75.7 to 93.6]
  B/Victoria//Day 28: number analyzed (Participants) | 0 | 63 | 67
  B/Victoria//Day 28 |  | 73.0 [60.3 to 83.4] | 79.1 [67.4 to 88.1]
  B/Victoria//Day 56: number analyzed (Participants) | 0 | 61 | 66
  B/Victoria//Day 56 |  | 91.8 [81.9 to 97.3] | 84.8 [73.9 to 92.5]

14. Secondary Outcome: Percentage of Participants With Any Post Dose Strain-specific Antibody Response
Description: Strain specific antibody response defined as >= 4-fold increase in HAI antibodies or >= 4-fold increase in neutralizing antibodies or >= 2-fold increase in IgA antibodies.
Time Frame: Days 28 and 56
Population: Immunogenicity population. B/Victoria strain was not included in the 'FluMist trivalent (2015-2016)' arm.
Measure: Number; unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 66 | 65 | 67
Percentage of participants
  A/H1N1/HAI response/Day 28: number analyzed (Participants) | 60 | 56 | 64
  A/H1N1/HAI response/Day 28 | 10.0 | 5.4 | 23.4
  A/H1N1/Microneutralization response/Day 28: number analyzed (Participants) | 60 | 56 | 63
  A/H1N1/Microneutralization response/Day 28 | 3.3 | 5.4 | 15.9
  A/H1N1/Nasal IgA response/Day 28: number analyzed (Participants) | 63 | 63 | 67
  A/H1N1/Nasal IgA response/Day 28 | 46.0 | 52.4 | 35.8
  A/H1N1/HAI response/Day 56: number analyzed (Participants) | 59 | 56 | 62
  A/H1N1/HAI response/Day 56 | 23.7 | 12.5 | 45.2
  A/H1N1/Microneutralization response/Day 56: number analyzed (Participants) | 59 | 56 | 60
  A/H1N1/Microneutralization response/Day 56 | 15.3 | 10.7 | 31.7
  A/H1N1/Nasal IgA response/Day 56: number analyzed (Participants) | 64 | 60 | 65
  A/H1N1/Nasal IgA response/Day 56 | 46.9 | 53.3 | 61.5
  A/H3N2/HAI response/Day 28: number analyzed (Participants) | 60 | 56 | 64
  A/H3N2/HAI response/Day 28 | 51.7 | 64.3 | 31.3
  A/H3N2/Microneutralization response/Day 28: number analyzed (Participants) | 60 | 56 | 63
  A/H3N2/Microneutralization response/Day 28 | 60.0 | 66.1 | 30.2
  A/H3N2/Nasal IgA response/Day 28: number analyzed (Participants) | 64 | 62 | 67
  A/H3N2/Nasal IgA response/Day 28 | 81.3 | 85.5 | 38.8
  A/H3N2/HAI response/Day 56: number analyzed (Participants) | 59 | 56 | 62
  A/H3N2/HAI response/Day 56 | 54.2 | 66.1 | 40.3
  A/H3N2/Microneutralization response/Day 56: number analyzed (Participants) | 59 | 56 | 60
  A/H3N2/Microneutralization response/Day 56 | 57.6 | 69.6 | 30.0
  A/H3N2/Nasal IgA response/Day 56: number analyzed (Participants) | 64 | 61 | 65
  A/H3N2/Nasal IgA response/Day 56 | 76.6 | 82.0 | 50.8
  B/Yamagata/HAI response/Day 28: number analyzed (Participants) | 60 | 56 | 64
  B/Yamagata/HAI response/Day 28 | 50.0 | 42.9 | 57.8
  B/Yamagata/Microneutralization response/Day 28: number analyzed (Participants) | 60 | 56 | 64
  B/Yamagata/Microneutralization response/Day 28 | 48.3 | 37.5 | 48.4
  B/Yamagata/Nasal IgA response/Day 28: number analyzed (Participants) | 64 | 63 | 67
  B/Yamagata/Nasal IgA response/Day 28 | 65.6 | 87.3 | 61.2
  B/Yamagata/HAI response/Day 56: number analyzed (Participants) | 60 | 56 | 62
  B/Yamagata/HAI response/Day 56 | 50.0 | 53.6 | 54.8
  B/Yamagata/Microneutralization response/Day 56: number analyzed (Participants) | 60 | 56 | 62
  B/Yamagata/Microneutralization response/Day 56 | 61.7 | 57.1 | 61.3
  B/Yamagata/Nasal IgA response/Day 56: number analyzed (Participants) | 64 | 61 | 66
  B/Yamagata/Nasal IgA response/Day 56 | 70.3 | 83.6 | 77.3
  B/Victoria/HAI response/Day 28: number analyzed (Participants) | 0 | 56 | 64
  B/Victoria/HAI response/Day 28 |  | 14.3 | 35.9
  B/Victoria/Microneutralization response/Day 28: number analyzed (Participants) | 0 | 56 | 63
  B/Victoria/Microneutralization response/Day 28 |  | 19.6 | 17.5
  B/Victoria/Nasal IgA response/Day 28: number analyzed (Participants) | 0 | 63 | 67
  B/Victoria/Nasal IgA response/Day 28 |  | 76.2 | 55.2
  B/Victoria/HAI response/Day 56: number analyzed (Participants) | 0 | 56 | 62
  B/Victoria/HAI response/Day 56 |  | 25.0 | 40.3
  B/Victoria/Microneutralization response/Day 56: number analyzed (Participants) | 0 | 56 | 60
  B/Victoria/Microneutralization response/Day 56 |  | 16.1 | 21.7
  B/Victoria/Nasal IgA response/Day 56: number analyzed (Participants) | 0 | 61 | 66
  B/Victoria/Nasal IgA response/Day 56 |  | 83.6 | 78.8

15. Secondary Outcome: Percentage of Participants With Any Solicited Symptoms
Description: Solicited symptoms included fever by any route (temperature >= 100.4 degrees Fahrenheit), runny/stuffy nose, sore throat, cough, headache, generalized muscle aches, lethargy or tiredness/weakness, and decreased appetite.
Time Frame: Day 1 through Day 14 after Dose 1 (Day 1 dose) and Dose 2 (Day 28 dose)
Population: ATP included all participants who received any investigational drug.
Measure: Number; unit: Percentage of participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 67 | 66 | 67
Percentage of participants
  Fever: Dose 1: number analyzed (Participants) | 67 | 65 | 67
  Fever: Dose 1 | 3.0 | 1.5 | 10.4
  Fever: Dose 2: number analyzed (Participants) | 63 | 61 | 63
  Fever: Dose 2 | 3.2 | 8.2 | 6.3
  Runny/Stuffy Nose: Dose 1: number analyzed (Participants) | 67 | 65 | 67
  Runny/Stuffy Nose: Dose 1 | 34.3 | 41.5 | 43.3
  Runny/Stuffy Nose: Dose 2: number analyzed (Participants) | 63 | 60 | 64
  Runny/Stuffy Nose: Dose 2 | 33.3 | 36.7 | 34.4
  Sore Throat: Dose 1: number analyzed (Participants) | 67 | 65 | 67
  Sore Throat: Dose 1 | 6.0 | 1.5 | 4.5
  Sore Throat: Dose 2: number analyzed (Participants) | 63 | 60 | 64
  Sore Throat: Dose 2 | 3.2 | 3.3 | 4.7
  Cough: Dose 1: number analyzed (Participants) | 67 | 65 | 67
  Cough: Dose 1 | 19.4 | 15.4 | 10.4
  Cough: Dose 2: number analyzed (Participants) | 63 | 60 | 64
  Cough: Dose 2 | 19.0 | 21.7 | 10.9
  Headache: Dose 1: number analyzed (Participants) | 67 | 65 | 67
  Headache: Dose 1 | 1.5 | 4.6 | 6.0
  Headache: Dose 2: number analyzed (Participants) | 63 | 60 | 64
  Headache: Dose 2 | 3.2 | 5.0 | 3.1
  Generalized Muscle Aches: Dose 1: number analyzed (Participants) | 67 | 65 | 67
  Generalized Muscle Aches: Dose 1 | 4.5 | 4.6 | 1.5
  Generalized Muscle Aches: Dose 2: number analyzed (Participants) | 63 | 60 | 64
  Generalized Muscle Aches: Dose 2 | 0.0 | 3.3 | 0.0
  Lethargy/Tiredness/Weakness: Dose 1: number analyzed (Participants) | 67 | 65 | 67
  Lethargy/Tiredness/Weakness: Dose 1 | 13.4 | 13.8 | 16.4
  Lethargy/Tiredness/Weakness: Dose 2: number analyzed (Participants) | 63 | 60 | 64
  Lethargy/Tiredness/Weakness: Dose 2 | 12.7 | 11.7 | 7.8
  Decreased Appetite: Dose 1: number analyzed (Participants) | 67 | 65 | 67
  Decreased Appetite: Dose 1 | 13.4 | 12.3 | 11.9
  Decreased Appetite: Dose 2: number analyzed (Participants) | 63 | 60 | 64
  Decreased Appetite: Dose 2 | 9.5 | 8.3 | 7.8

16. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An Adverse Event (AE) is any unfavourable and unintended sign, symptoms, or diseases temporally associated with use of study drug, whether or not considered related to study drug. A serious adverse event (SAE) is an AE that results in death, initial or prolonged inpatient hospitalization, life-threatening, persistent or significant disability/incapacity, congenital anomaly/birth defect, or an important medical event. TEAEs and TESAEs are defined as AEs and SAEs present at baseline that worsened in intensity after administration of study drug, or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through Day 28 after Dose 1 (Day 1 dose) and Dose 2 (Day 28 dose)
Population: ATP included all participants who received any investigational drug.
Measure: Count of Participants; unit: Participants
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
Number analyzed (Participants) | 67 | 66 | 67
Participants
  TEAEs | 29 | 31 | 34
  TESAEs | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 through Day 28 after Dose 1 (Day 1 dose) and Dose 2 (Day 28 dose)
Description: ATP included all participants who received any investigational drug.
Arm/Group | FluMist Trivalent (2015-2016) | FluMist Quadrivalent (2015-2016) | FluMist Quadrivalent (2017-2018)
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/66 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/66 | 0/67
Other Adverse Events (participants affected / at risk) | 29/67 | 31/66 | 34/67
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FluMist Trivalent (2015-2016) (N=67) | FluMist Quadrivalent (2015-2016) (N=66) | FluMist Quadrivalent (2017-2018) (N=67)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Eye oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 5 (5) | 4 (5)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 5 (6) | 4 (5)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Developmental delay (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 7 (7) | 2 (2)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Croup infectious (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 3 (4) | 1 (1) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 1 (1) | 3 (4)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2) | 2 (2)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radial head dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 4 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7) | 9 (9)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/01/NCT03143101/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT03143101/SAP_001.pdf